CLINICAL TRIAL: NCT05095064
Title: Retrospective Study on the Efficacy and Tolerability of Liposomal irinotecanN (MM398, PEP02, Onivyde) for the Treatment of Pancreatic Adenocarcinoma.
Brief Title: Retrospective Study on the Efficacy and Tolerability of Liposomal Irinotecan
Acronym: NALIRI
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Universitair Ziekenhuis Brussel (Other); AZ Nikolaas (Other); General Hospital Groeninge (Other); University Hospital St Luc, Brussels (Other); ASZ Aalst (Other); Erasme University Hospital (Other); Centre Hospitalier Universitaire de Liege (Other); OLVZ Ziekenhuis Aalst (Unknown)
Responsible Party: Sponsor
Other Study IDs: EDGE 001385
Record Dates: First submitted 2021-09-21; First posted 2021-10-27 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2021-10

CONDITIONS: Metastatic Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — irinotecan sucrosofate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Onivyde® + 5-FULV — Nanoliposomal irinotecan (Onivyde®) in combination with 5-fluorouracil and leucovorin (5-FU/LV)
  Other Names: Nanoliposomal irinotecan

SUMMARY:
The aim of this retrospective study is to confirm the efficacy and safety results obtained in the NAPOLI-1-study, when Onivyde® in combination with 5-FU/LV is used in real-life practice in Belgium. The data needed to do so will be obtained using information that is routinely collected as part of patient's medical care.

DETAILED DESCRIPTION:
Patients with pancreatic cancer have a poor prognosis with a 5-years survival of only 1-2%. This arises from the fact that it is typically diagnosed late, when curative resection is impossible. These patients are thus restricted to chemotherapy, with gemcitabine-based therapies being the standard of care for patients with locally advanced or metastatic pancreatic ductal adenocarcinoma (mPDAC). However, even after second or subsequent lines of therapy, disease progression is inevitable. Therefore, the need for new treatment options is high. Recently, the advantage of using nanoliposomal irinotecan (Onivyde®) in combination with 5-fluorouracil and leucovorin (5-FU/LV) over the use of 5-FU/LV alone was demonstrated in a phase-3 randomized clinical trial (NAPOLI-1 trial). As this study showed significant improvement on overall survival, progression-free survival, time to treatment failure, overall response rate and tumor marker CA19-9 response, on October 14 2016 this therapy was approved by the EMA to be used for patients with mPDAC previously treated with gemcitabine-based therapy.

While randomized clinical trials, like the NAPOLI-1 trial, are considered the reference standard for comparing the efficacy and safety of treatments, these studies do not always reflect the everyday clinical practice. Therefore, the aim of this study is to evaluate the efficacy and safety of Onivyde® in real-life practice in Belgium. This information would be very valuable to determine the value of the drug and improve the knowledge of the actual use of Onivyde® after marketing authorization.

ELIGIBILITY:
Inclusion Criteria:

* Patient has diagnosis of pancreatic adenocarcinoma with documented metastatic disease.
* Patient progressed after gemcitabine-based therapy.
* Patient received at least one treatment cycle with Onivyde® + 5-FU/LV 5FU in the context of post-gemcitabine based therapy of mPDAC.

Exclusion Criteria:

* Patient has not received at least one treatment cycle with Onivyde® + 5-FU/LV.
* Previous irinotecan-based therapy in metastatic setting.
* Patientstarted the treatment with Onivyde® + 5-FU/LV after 01/04/2021

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Metastatic pancreatic ductal adenocarcinoma
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
The overall survival (OS) from start of treatment with Onivyde® + 5-FU/LV | 03/2022
  All this info is retrospectively obtained from the patients medical fistory. Data analysis is forseen to be finished 03/2022.

SECONDARY OUTCOMES:
Survival rate at 2, 4, 6, 8, 10 months from the start of treatment with Onivyde® + 5-FU/LV | 03/2022
  All this info is retrospectively obtained from the patients medical history. Data analysis is forseen to be finished 03/2022.
Progression-free survival (PFS) from the start of Onivyde® + 5-FU/LV treatment | 03/2022
  All this info is retrospectively obtained from the patients medical history. Data analysis is forseen to be finished 03/2022.
Disease control rate of patients from the start of treatment with Onivyde® + 5-FU/LV | 03/2022
  All this info is retrospectively obtained from the patients medical history. Data analysis is forseen to be finished 03/2022.
Change in baseline performance status of the patient after Onivyde® + 5-FU/LV treatment | 03/2022
  All this info is retrospectively obtained from the patients medical history. Data analysis is forseen to be finished 03/2022.
The OS from the date of diagnosis of metastatic disease | 03/2022
  All this info is retrospectively obtained from the patients medical history. Data analysis is forseen to be finished 03/2022.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Peeters, Principal Investigator — University Hospital, Antwerp
Locations (1):
- Antwerp University Hosptital, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Verbruggen L, Verheggen L, Vanhoutte G, Loly C, Lybaert W, Borbath I, Vergauwe P, Hendrickx K, Debeuckelaere C, de Haar-Holleman A, Van Laethem JL, Peeters M. A real-world analysis on the efficacy and tolerability of liposomal irinotecan plus 5-fluorouracil and folinic acid in metastatic pancreatic ductal adenocarcinoma in Belgium. Ther Adv Med Oncol. 2023 Aug 18;15:17588359231181500. doi: 10.1177/17588359231181500. eCollection 2023. PMID 37600936